CLINICAL TRIAL: NCT00478959
Title: Phase II Study of Lenalidomide for the Treatment of Relapsed or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-HL
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Hodgkin Disease
Keywords: Lenalidomide; Revlimid; Hodgkin's; Hodgkin; Hodgkin's Lymphoma; Hodgkin's Disease; Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide given as a daily oral dose of 25 mg on days 1 - 21 followed by 7 days of no therapy of a 28 day cycle in the treatment of a population with relapsed or refractory Hodgkin's lymphoma.
  Interventions: Drug: Lenalidomide (Revlimid®)

INTERVENTIONS:
Drug: Lenalidomide (Revlimid®) — 25mg PO daily for 21 out of 28days per cycle
  Other Names: Revlimid

SUMMARY:
This is a single-arm, open-label Phase II study evaluating the activity of Lenalidomide in patients with relapsed or refractory Hodgkin's lymphoma.

DETAILED DESCRIPTION:
While the results of primary therapy for Hodgkin's lymphoma are generally excellent, between 10-20% of patients with advanced stage disease will not enter a complete remission (CR) and between 20-30% of patients will relapse after completion of treatment. Salvage chemotherapy followed by high dose chemotherapy and autologous stem cell transplantation (ASCT) has become the treatment of choice in patients with relapsed or initially chemotherapy-refractory disease.

Although high dose chemotherapy remains a curative option for the treatment of relapsed or chemotherapy-refractory Hodgkin's lymphoma, up to 50% of patients will ultimately recur post-stem cell transplant and will require further treatment.

Thalidomide is an agent that has anti-inflammatory, immunomodulatory and anti-angiogenic properties. Thalidomide has been shown to have activity in a number of solid and hematologic malignancies, and has demonstrated effectiveness in the treatment of refractory multiple myeloma. A dose escalation study of single-agent thalidomide has been performed in heavily pre-treated patients in which two Hodgkin's patients were enrolled and did not respond to treatment. Based on the NCI experience with vinblastine, we initiated a phase II trial examining the combination of thalidomide and vinblastine in patients who were being treated palliatively for Hodgkin's lymphoma. In a heavily pre-treated group of patients (70% of cases having relapsed post-ASCT), a response rate of 40% to the combination was noted with median duration of response of over nine months.

Lenalidomide (Revlimid®) is a thalidomide derivative and the first-in-class novel immunomodulatory agent that has more potent activity as well as a more favourable toxicity profile than the parent compound. Based on the alterations demonstrated in various cytokines and angiogenic markers in patients with Hodgkin's lymphoma, we feel that Lenalidomide's immunomodulatory and anti-angiogenic effects make this an ideal drug to study in this lymphoma. This will be the first study to assess Lenalidomide in patients with Hodgkin's lymphoma.This is a single arm, open-label phase II multi-centre study evaluating the single agent activity of Lenalidomide in relapsed or refractory Hodgkin's lymphoma. The primary endpoint is objective response rate (CR + CRu + PR) as determined by International Workshop Criteria.

Initial treatment will consist of lenalidomide 25 mg PO daily given for 21 consecutive days (days 1 - 21), with seven days off on a 28 day cycle.Patients with PR, CR or CRu, may continue on therapy for 2 cycles past best response.Patients with PD at any time or those with evidence of SD after cycle 4 of monotherapy will be eligible to receive treatment with dexamethasone 40 mg PO daily on days 1 - 4 and 15 - 18 of a 28 day cycle while continuing protocol treatment if they continue to meet the criteria of continuation on therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Hodgkin's lymphoma that is relapsed or refractory (repeat biopsy is not mandatory) and is no longer eligible for curative treatment
* </=3 prior chemotherapy regimens (in patients without a prior ASCT)
* Patients with disease progression after ASCT will be eligible if they have received </= 1 additional chemotherapy regimen post-ASCT
* ECOG Performance Status 0-2
* Adequate hematological function:

  * Absolute granulocyte count > 1.0 x 10 to the 9/L
  * Platelet count > 75 x 10 to the 9/L
* Adequate renal and hepatic functions:

  * Serum creatinine < 1.25 x UNL or a calculated creatinine clearance > 50 mL/min
  * Serum bilirubin < 1.5 x UNL and AST/ALT < 3 x UNL
* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL 10 - 14 days prior to therapy and repeated within 24 hours of starting study drug and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. Women must also agree to ongoing pregnancy testing. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential. (See Appendix B Pregnancy Testing Guidelines and Acceptable Birth Control Methods.)
* Able to take aspirin (325 mg daily) as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin)
* Written Informed Consent must be given according to ICH/GCP and national/local regulations

Exclusion Criteria

* Prior treatment with Lenalidomide or Thalidomide
* Use of any other experimental therapy within the 28 days prior to baseline assessment
* Known infection with Human Immunodeficiency Virus (HIV), Hepatitis B or C
* Pregnant or Lactating women
* Other significant medical problems such as uncontrolled hypertension, uncontrolled psychiatric symptoms disorders, serious infections, active peptic ulcer disease, or any other medical conditions that might be aggravated by treatment
* Second malignancy in the past five years with the exception of adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix or breast
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.
* Concurrent use of other anti-cancer agents or treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To assess the response rate (CR + CRu + PR) of Lenalidomide given as a daily oral dose of 25 mg on days 1 - 21 followed by 7 days of no therapy of a 28 day cycle in the treatment of a population with relapsed or refractory Hodgkin's lymphoma | CT scans performed every two months while on therapy

CONTACTS AND LOCATIONS:
Overall Officials: John Kuruvilla, Principal Investigator — Princess Margaret Hospital, Canada